CLINICAL TRIAL: NCT03408431
Title: Effect of the Neck Extension on Blind Intubation Via Ambu® AuraGain™ Laryngeal Mask: a Randomized Controlled Trial
Brief Title: Effect of the Neck Extension on Blind Intubation Via Ambu® AuraGain™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-1709-123-890
Record Dates: First submitted 2018-01-10; First posted 2018-01-24 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Intubation; Difficult or Failed; Intubation Complication

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group E (Experimental): After the placement of Ambu® AuraGain™, blind intubation will be performed in patients assigned group E with neck extension positioning.
  Interventions: Device: Ambu® AuraGain™; Procedure: neck extension
- Group C (Active Comparator): After the placement of Ambu® AuraGain™, blind intubation will be performed in patients assigned group E with neutral head and neck position.
  Interventions: Device: Ambu® AuraGain™

INTERVENTIONS:
Device: Ambu® AuraGain™ — Ambu® AuraGain™ laryngeal mask will be placed first, and then, a lubricated endotracheal tube will be gently intubated through the laryngeal mask under each position according to the assigned group.
Procedure: neck extension — Patients' neck will be maximally extended (~60°) during blind intubation.
  Arms: Group E

SUMMARY:
In a previous study, NCT03147469, the investigators found that the vocal cords were more easily visualized by fiberoptic bronchoscopy with neck extension positioning. On the basis of this finding, the investigators are going to conduct a randomized controlled trial to evaluate the effect of neck extension on the success rate of blind intubation through laryngeal mask.

Participants undergoing general anesthesia will be randomly assigned to group E (with neck extension) or group C (with neutral position). Ambu® AuraGain™ laryngeal mask will be placed first, and then, a lubricated endotracheal tube will be gently intubated through the laryngeal mask. The participants will be mechanically ventilated with an endotracheal tube if blind intubation succeed. Blind intubation will be performed with a maximum of two attempts. If all attempts failed, the laryngeal mask will be removed and the tube will be intubated using a direct laryngoscopy.

The primary outcome of this study is the success rate of blind intubation within a first attempt. Secondary outcomes included overall success rate of blind intubation within a maximum of two attempts, time for blind intubation, the incidence of postoperative hoarseness, cough, and sore throat, and any obvious complications related to airway management such as bleeding, airway trauma, dental fracture, aspiration, or bronchospasm.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing general anesthesia with endotracheal intubation

Exclusion Criteria:

* Emergency operation
* History of esophageal, oropharyngeal, or laryngeal disease
* History of cervical spine surgery
* Insufficient NPO time
* Loosening teeth
* Mouth opening less than 2cm

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Success rate in first attempt | In a first attempt for blind intubation, an average of 30 seconds
  Successful blind intubation in a first attempt

SECONDARY OUTCOMES:
Overall success rate | In a maximum of two attempts for blind intubation, an average of 60 seconds
  Successful blind intubation within a maximum of two attempts
Time for blind intubation | In a maximum of two attempts for blind intubation, an average of 60 seconds
  Time between insertion of an endotracheal tube within the laryngeal mask and detection of end-tidal CO2 from the tube
Postoperative hoarseness | 24 hours after extubation
  The incidence of postoperative hoarseness
Postoperative cough | 24 hours after extubation
  The incidence of postoperative cough
Postoperative sore throat | 24 hours after extubation
  The incidence of postoperative sore throat

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yoo S, Park SK, Kim WH, Hur M, Bahk JH, Lim YJ, Kim JT. The effect of neck extension on success rate of blind intubation through Ambu(R) AuraGain laryngeal mask: a randomized clinical trial. Can J Anaesth. 2019 Jun;66(6):639-647. doi: 10.1007/s12630-019-01353-4. Epub 2019 Mar 27. PMID 30919236